CLINICAL TRIAL: NCT04318691
Title: Netosis in Mechanically Ventilated ICU Patients in Determination of Respiratory Infection Severity
Brief Title: Netosis in Determination of Respiratory Infection Severity
Acronym: NETMINDERS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00217-32
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Infection
Keywords: acute respiratory distress syndrome; adult ICU; neutrophil extracellular traps (NETs); Netosis; neutrophils; mechanical ventilation; pneumonia
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Distress Syndrome; Pneumonia | interventions — Blood Specimen Collection; Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- acute respiratory failure group: 60 patients under mechanical ventilation admitted to the intensive care unit for acute respiratory failure
  Interventions: Biological: Blood sampling; Procedure: Bronchoalveolar lavage
- vascular surgery control group: 10 control patients admitted to the ICU after a planned vascular surgery
  Interventions: Biological: Blood sampling
- Healthy volunteers group: 10 healthy subjects.
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood sampling at baseline and at day-3 (10 ml, EDTA tube), test of NETs.
Procedure: Bronchoalveolar lavage — Bronchoalveolar lavage at admission to the ICU with analysis of cytological, bacteriological, viral and anatomopathological, and test of NETs.
  Groups: acute respiratory failure group

SUMMARY:
The study aims to evaluate the prognostic value of alveolar and blood NETosis in patients under mechanical ventilation and treated for an acute low-respiratory tract infection. The main outcome is the occurrence of an acute respiratory distress syndrome (ARDS) according to the Berlin definition.

DETAILED DESCRIPTION:
Neutrophils are the first line of defense against infectious injury. Among the numerous mechanisms involving the immune system, neutrophil extracellular traps (NETs) have been recently described as an additional way neutrophils are able to use to fight against bacteria. NETs are made of DNA and antimicrobial proteins. In the other hand, NETs promote coagulation and may contribute to evolution of severe pneumonia into acute respiratory distress syndrome.

The secondary objectives of the study include the research of the relation between blood NETosis and alveolar NETosis with:

* the documentation of invasive pulmonary infection based on microbiological analysis criteria (which would be bacteria or viral) of LBA at admission to ICU;
* the diagnosis value of usually used biomarkers: procalcitonin and C-reactive protein;
* marbrure score at admission to ICU;
* arterial lactatemia;
* scores of gravity at admission IGSII and SOFA;
* all-cause mortality at day-28;
* duration of mechanical ventilation at day-28;
* duration of amines at day-28;
* developement of hemodynamic failure;
* developement of pulmonary circulatory failure.

The study will include 1) 60 patients under mechanical ventilation admitted to the intensive care unit for acute respiratory failure, 2) 10 control patients admitted to the ICU after a planned vascular surgery and 3) 10 healthy subjects.

ELIGIBILITY:
Inclusion criteria:

A/ For all subjets:

* Be >/= 18 years of age on day of signing informed consent;
* Affiliated to the french social security - welfare system in France.

B/ Inclusion criteria for acute respiratory failure patients:

admitted to the ICU for acute respiratory failure requiring mechanical ventilation within the first 24 hours after admission and suspected to suffer from an infectious pneumonia, according to the following criteria:

* recent fever;
* acute respiratory failure signs (dyspnea, polypnea > 30 cycles/min, hypoxemia PaO2<65 mmHg);
* pulmonary focal signs of auscultation;
* evocative signs in chest radiography or chest TDM.

C/ Inclusion criteria for control patients:

- admitted to the ICU for post-operative management of vascular surgery.

Exclusion Criteria:

A/ For all subjets:

* pregnancy,
* nosocomial pneumonia,
* no social health insurance,
* neutropenia of any cause;
* patient refusal.

B/ Exclusion criteria for acute respiratory failure patients:

- no mechanical ventilation within the first 24 hours after admission to the ICU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adult ICU patients under mechanical ventilation with suspected lower-respiratory tract infection;
  * Adult ICU patients followed vascular surgical intervention;
  * Healthy Volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Acute respiratory distress syndrome occurrence | at day-7
  Acute respiratory distress syndrome occurrence according to the Berlin definition within the first 7 days after ICU admission

SECONDARY OUTCOMES:
Mortality | At day-28
  Vital statue of patient
Duration of mechanical ventilation | At day-28
  Duration of mechanical ventilation: number of days without mechanical ventilation.
IGSII score | At admission to ICU
  IGSII score
SOFA score | At admission to ICU
  SOFA score
Hemodynamic failure | At day-28
  Development of a hemodynamic failure
Pulmonary circulation failure | At day-28
  Development of a pulmonary circulation failure (acute pulmonary heart disease, right ventricle failure)

CONTACTS AND LOCATIONS:
Overall Officials: Edouard JULLIEN, MD, Principal Investigator — Service de médecine intensive réanimation, Hôpital Ambroise Paré, APHP; Guillaume Geri, MD, PhD, Study Director — Service de médecine intensive réanimation, Hôpital Ambroise Paré, APHP
Locations (1):
- Service de médecine intensive réanimation, Hôpital Ambroise Paré, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No